CLINICAL TRIAL: NCT05935631
Title: Feasibility, Acceptability and Directional Signal Effect on Blood Folate Levels of Iodized Salt Fortified With Folic Acid: Clinical Study
Acronym: FASALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Anastasia Arynchyna, Clinical Research Manager/ DrPH student, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 300009522
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neural Tube Defects; Folic Acid Deficiency; Fortification
Keywords: Serum folate
MeSH Terms: conditions — Neural Tube Defects; Folic Acid Deficiency | interventions — Salts; Folic Acid; Iodine

STUDY DESIGN:
Intervention Model Description: Pre-test and post-test of serum folate levels after using salt with folic acid in the same group of women, each serving as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salt with folic acid and iodine (Experimental): Intervention is intake of double fortified salt with folic acid and iodine (DFS). We will ask the participants to substitute their current salt with the study saltshaker and use it when preparing food or when eating out. We estimate minimum daily intake from salt consumption by participants will be 200 micrograms (µg) of folic acid per serving. Serving is 2g of salt. Participants will be given portion suggestions: 1/2 teaspoon or 2-3 pinches or 8-10 shakes/5 times a day. Containers (125g) will be weighted at the beginning and end of 1 month. We will ask each day if woman cooked/used the salt for herself only or to list number of people each day. Participants will also agree to complete either daily paper salt log. A commercially available salt that is fortified with folic acid has been provided by AlpenJodSalz produced by Sudwestdeutsche Salzwerk. For 30 participants, we will need 30 containers.
  Interventions: Dietary Supplement: Salt with folic acid and iodine

INTERVENTIONS:
Dietary Supplement: Salt with folic acid and iodine — Assess serum and RBC folate levels in women at baseline and 1 month after ingesting salt with folic acid

SUMMARY:
Aim 1: Assess directional signal of effect of fortified salt with folic acid and iodine on blood serum folate levels.

It will be accomplished by feasibility pre-test/post-test clinical study by estimating mean and variability of serum blood folate levels effects of folic acid fortified salt.

Hypothesis: Fortified salt with folic acid and iodine will increase serum blood folate levels from baseline by month 1.

Aim 2: Assess feasibility and acceptability of salt fortified with folic acid and iodine.

Feasibility will be measured by 1) subjects' refusal rate of consent by 30 subjects during 6-month enrollment period; 2) method of determining salt consumption (weighting the saltshaker pre and post); 3) completion rates of study protocols from baseline to follow up. Hypothesis 1a: Completion of all blood draw visits will be 90-100%.

Acceptability will be measured by 1) completion rate of daily salt logs; 2) consumption of salt by weighting saltshakers; 3) attitude towards taste and color difference. Hypothesis 1b: Completion rate (90-100%) of daily salt logs will range from 90-100% of participants and 2) consumption of salt will range from 90-100% of participants.

Dietary surveys will be employed to document dietary habits and estimated daily FA intake in the sample population. Feasibility and acceptability of dietary surveys will be measured by willingness to answer survey questions. Hypothesis 1c: Completion rate of dietary surveys will range 90-100%.

ELIGIBILITY:
Inclusion Criteria:

* women
* consumes salt

Exclusion Criteria:

* pregnant or intends to become pregnant in next 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are focusing on women specifically as we looking at maternal blood folate levels prior to potential pregnancy
Enrollment: 32 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Serum blood folate levels | One month
  Change in serum blood folate levels from baseline to one month

SECONDARY OUTCOMES:
Number of participants who are enrolled in the study | one month
  Feasibility of enrollment: number of participants who are enrolled in the study
Change in weight of salt shakers (in grams) | one month
  Acceptability of salt with folic acid and iodine by the participants through weighting salt shackers before and after and calculating amount of salt ingested.
Percent of participants who completed all study visits | one month
  Percent of participants who completed all study visits
Measure of effect salt with folic acid had on taste of food using Likert scale | one month
  Did using this salt negatively affect the taste of your food overall? It is measured on Likert scale (1- strongly disagree, 5 strongly agree)
Measure of whether the color of salt negatively affect their desire to use it daily using Likert Scale | one month
  Did the color of salt negatively affect your desire to use it daily? It is measured on Likert scale (1- strongly disagree, 5 strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Arynchyna-Smith, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
If another investigator has a valid research question and hypothesis that fits in with the study sample, we will consider sharing de-identified dataset. Participants have consented to share their de-identified data with future researchers.

REFERENCES:
- [Background] Kancherla V, Wagh K, Pachon H, Oakley GP Jr. A 2019 global update on folic acid-preventable spina bifida and anencephaly. Birth Defects Res. 2021 Jan 1;113(1):77-89. doi: 10.1002/bdr2.1835. Epub 2020 Oct 30. PMID 33124747
- [Background] Kancherla V, Tsang B, Wagh K, Dixon M, Oakley GP Jr. Modeling shows high potential of folic acid-fortified salt to accelerate global prevention of major neural tube defects. Birth Defects Res. 2020 Nov;112(18):1461-1474. doi: 10.1002/bdr2.1769. Epub 2020 Aug 1. PMID 32738033
- [Background] Blencowe H, Kancherla V, Moorthie S, Darlison MW, Modell B. Estimates of global and regional prevalence of neural tube defects for 2015: a systematic analysis. Ann N Y Acad Sci. 2018 Feb;1414(1):31-46. doi: 10.1111/nyas.13548. Epub 2018 Jan 24. PMID 29363759
- [Background] Allen R, James A, Sankaran S. Trends in termination of pregnancy for neural tube defects in England and Wales from 2007 to 2017: Observational prospective study. Prenat Diagn. 2021 Dec;41(13):1624-1633. doi: 10.1002/pd.6060. Epub 2021 Oct 26. PMID 34671992
- [Background] Lynberg MC, Khoury MJ. Contribution of birth defects to infant mortality among racial/ethnic minority groups, United States, 1983. MMWR CDC Surveill Summ. 1990 Jul;39(3):1-12. PMID 2115106
- [Background] Hopson B; MSHA; Alford EN, Zimmerman K, Blount JP, Rocque BG. Development of an evidence-based individualized transition plan for spina bifida. Neurosurg Focus. 2019 Oct 1;47(4):E17. doi: 10.3171/2019.7.FOCUS19425. PMID 31574471
- [Background] Crider KS, Devine O, Hao L, Dowling NF, Li S, Molloy AM, Li Z, Zhu J, Berry RJ. Population red blood cell folate concentrations for prevention of neural tube defects: Bayesian model. BMJ. 2014 Jul 29;349:g4554. doi: 10.1136/bmj.g4554. PMID 25073783
- [Background] Estevez-Ordonez D, Davis MC, Hopson B; MSHA; Arynchyna A, Rocque BG, Fieggen G, Rosseau G, Oakley G; MSPM; Blount JP. Reducing inequities in preventable neural tube defects: the critical and underutilized role of neurosurgical advocacy for folate fortification. Neurosurg Focus. 2018 Oct;45(4):E20. doi: 10.3171/2018.7.FOCUS18231. PMID 30269587
- [Background] Oumer M, Tazebew A, Silamsaw M. Birth prevalence of neural tube defects and associated risk factors in Africa: a systematic review and meta-analysis. BMC Pediatr. 2021 Apr 21;21(1):190. doi: 10.1186/s12887-021-02653-9. PMID 33882899
- [Background] Williams J, Mai CT, Mulinare J, Isenburg J, Flood TJ, Ethen M, Frohnert B, Kirby RS; Centers for Disease Control and Prevention. Updated estimates of neural tube defects prevented by mandatory folic Acid fortification - United States, 1995-2011. MMWR Morb Mortal Wkly Rep. 2015 Jan 16;64(1):1-5. PMID 25590678
- [Background] Kancherla V, Wagh K, Priyadarshini P, Pachon H, Oakley GP Jr. A global update on the status of prevention of folic acid-preventable spina bifida and anencephaly in year 2020: 30-Year anniversary of gaining knowledge about folic acid's prevention potential for neural tube defects. Birth Defects Res. 2022 Dec 1;114(20):1392-1403. doi: 10.1002/bdr2.2115. Epub 2022 Nov 7. PMID 36345648
- [Background] Wang A, Rose CE, Qi YP, Williams JL, Pfeiffer CM, Crider KS. Impact of Voluntary Folic Acid Fortification of Corn Masa Flour on RBC Folate Concentrations in the U.S. (NHANES 2011-2018). Nutrients. 2021 Apr 16;13(4):1325. doi: 10.3390/nu13041325. PMID 33923768
- [Background] Fan L, Meng F, Sun Q, Zhai Y, Liu P. Assessment of Sustainable Elimination Criteria for Iodine Deficiency Disorders Recommended by International Organizations. Front Nutr. 2022 Apr 13;9:852398. doi: 10.3389/fnut.2022.852398. eCollection 2022. PMID 35495946
- [Background] Liu T, Li Y, Teng D, Shi X, Yan L, Yang J, Yao Y, Ye Z, Ba J, Chen B, Du J, He L, Lai X, Teng X, Li Y, Chi H, Liao E, Liu C, Liu L, Qin G, Qin Y, Quan H, Shi B, Sun H, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yang L, Zhang Q, Zhang L, Zhu J, Zhu M, Shan Z, Teng W. The Characteristics of Iodine Nutrition Status in China After 20 Years of Universal Salt Iodization: An Epidemiology Study Covering 31 Provinces. Thyroid. 2021 Dec;31(12):1858-1867. doi: 10.1089/thy.2021.0301. Epub 2021 Dec 2. PMID 34806437
- [Background] Mokhort T, Petrenko S, Leushev B, Fedorenko E, Kolomiets N, Mokhort A. Assessment of iodine status among school age children and pregnant women of Belarus in 2017-2018. Clinical and experimental thyroidology. 11/13 2018;14doi:10.14341/ket9732
- [Background] Prevention of neural tube defects: results of the Medical Research Council Vitamin Study. MRC Vitamin Study Research Group. Lancet. 1991 Jul 20;338(8760):131-7. PMID 1677062
- [Background] Chen MY, Rose CE, Qi YP, Williams JL, Yeung LF, Berry RJ, Hao L, Cannon MJ, Crider KS. Defining the plasma folate concentration associated with the red blood cell folate concentration threshold for optimal neural tube defects prevention: a population-based, randomized trial of folic acid supplementation. Am J Clin Nutr. 2019 May 1;109(5):1452-1461. doi: 10.1093/ajcn/nqz027. PMID 31005964
- [Background] Eldridge C, Bandlamuri S, Andrews JG, Galindo MK, Contreras D, Flood TJ, Rice S. Postfolate spina bifida lesion level change. Birth Defects Res. 2018 Jul 3;110(11):949-955. doi: 10.1002/bdr2.1221. Epub 2018 Mar 25. PMID 29575817
- [Background] McDowell MA, Lacher DA, Pfeiffer CM, Mulinare J, Picciano MF, Rader JI, Yetley EA, Kennedy-Stephenson J, Johnson CL. Blood folate levels: the latest NHANES results. NCHS Data Brief. 2008 May;(6):1-8. PMID 19389320
- [Background] Pfeiffer CM, Sternberg MR, Zhang M, Fazili Z, Storandt RJ, Crider KS, Yamini S, Gahche JJ, Juan W, Wang CY, Potischman N, Williams J, LaVoie DJ. Folate status in the US population 20 y after the introduction of folic acid fortification. Am J Clin Nutr. 2019 Nov 1;110(5):1088-1097. doi: 10.1093/ajcn/nqz184. PMID 31504109
- [Background] Hopson B, Shamblin I, Zimmerman K, Rocque B, Salehani A, Blount JP. Scope of care in the first four years of life for individuals born with myelomeningocele: A single institution experience1. J Pediatr Rehabil Med. 2021;14(4):667-673. doi: 10.3233/PRM-200803. PMID 34864701
- [Background] Rocque BG, Bishop ER, Scogin MA, Hopson BD, Arynchyna AA, Boddiford CJ, Shannon CN, Blount JP. Assessing health-related quality of life in children with spina bifida. J Neurosurg Pediatr. 2015 Feb;15(2):144-9. doi: 10.3171/2014.10.PEDS1441. Epub 2014 Nov 21. PMID 25415252
- [Background] Mai CT, Evans J, Alverson CJ, Yue X, Flood T, Arnold K, Nestoridi E, Denson L, Adisa O, Moore CA, Nance A, Zielke K, Rice S, Shan X, Dean JH, Ethen M, Hansen B, Isenburg J, Kirby RS. Changes in Spina Bifida Lesion Level after Folic Acid Fortification in the US. J Pediatr. 2022 Oct;249:59-66.e1. doi: 10.1016/j.jpeds.2022.06.023. Epub 2022 Jun 27. PMID 35772508
- [Background] Mai CT, Isenburg J, Langlois PH, Alverson CJ, Gilboa SM, Rickard R, Canfield MA, Anjohrin SB, Lupo PJ, Jackson DR, Stallings EB, Scheuerle AE, Kirby RS; National Birth Defects Prevention Network. Population-based birth defects data in the United States, 2008 to 2012: Presentation of state-specific data and descriptive brief on variability of prevalence. Birth Defects Res A Clin Mol Teratol. 2015 Nov;103(11):972-93. doi: 10.1002/bdra.23461. No abstract available. PMID 26611917
- [Background] Grosse SD, Berry RJ, Mick Tilford J, Kucik JE, Waitzman NJ. Retrospective Assessment of Cost Savings From Prevention: Folic Acid Fortification and Spina Bifida in the U.S. Am J Prev Med. 2016 May;50(5 Suppl 1):S74-S80. doi: 10.1016/j.amepre.2015.10.012. Epub 2016 Jan 11. PMID 26790341
- [Background] McGee EJT, Sangakkara AR, Diosady LL. Double fortification of salt with folic acid and iodine. Journal of Food Engineering. 2017/04/01/ 2017;198:72-80. doi:https://doi.org/10.1016/j.jfoodeng.2016.11.019
- [Background] Modupe O, Krishnaswamy K, Diosady LL. Technology for Triple Fortification of Salt with Folic Acid, Iron, and Iodine. J Food Sci. 2019 Sep;84(9):2499-2506. doi: 10.1111/1750-3841.14730. Epub 2019 Aug 8. PMID 31393020
- [Background] Modupe O, Siddiqui J, Jonnalagadda A, Diosady LL. Folic acid fortification of double fortified salt. Sci Rep. 2021 Jul 15;11(1):14561. doi: 10.1038/s41598-021-93194-9. PMID 34267239
- [Background] Li YO, Diosady LL, Wesley AS. Folic acid fortification through existing fortified foods: iodized salt and vitamin A-fortified sugar. Food Nutr Bull. 2011 Mar;32(1):35-41. doi: 10.1177/156482651103200104. PMID 21560462
- [Background] Puri S, Rekhi TK, Thomas T, Jadhav MH, Mannar V, Diosady LL. Sensory Trial of Quintuple Fortified Salt-Salt Fortified With Iodine, Iron, Folic Acid, Vitamin B12, and Zinc-Among Consumers in New Delhi, India. Food Nutr Bull. 2022 Sep;43(3):340-350. doi: 10.1177/03795721221078361. Epub 2022 May 8. PMID 35531896
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Exchange GFD. Dashboard: Country Fortification. 2022. https://fortificationdata.org/country-fortification-dashboard/?alpha3_code=USA&lang=en
- [Background] Powles J, Fahimi S, Micha R, Khatibzadeh S, Shi P, Ezzati M, Engell RE, Lim SS, Danaei G, Mozaffarian D; Global Burden of Diseases Nutrition and Chronic Diseases Expert Group (NutriCoDE). Global, regional and national sodium intakes in 1990 and 2010: a systematic analysis of 24 h urinary sodium excretion and dietary surveys worldwide. BMJ Open. 2013 Dec 23;3(12):e003733. doi: 10.1136/bmjopen-2013-003733. PMID 24366578
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201